CLINICAL TRIAL: NCT03556345
Title: A Multicenter, Open Label，Single Arm，Phase II Study to Evaluate the Effect and Safety of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection in HER2 Overexpressing Local Advanced or Metastatic Gastric Cancer
Brief Title: A Study of RC48-ADC in Local Advanced or Metastatic Gastric Cancer Subjects With the Overexpression of HER2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C008
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Gastric Cancer; HER2 Overexpressing Gastric Carcinoma
Keywords: RC48-ADC; HER2 overexpression; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): Participants will receive RC48-ADC every 2 weeks (Q2W) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — 2.5 mg/kg IV every 2 weeks
  Other Names: Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC in local advanced or metastatic gastric patients with the overexpression of HER2.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years and ≤ 80 years.
* Predicted survival ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.
* Adequate organ function.
* Have had progression or intolerance following receipt of at least two systemic chemotherapy for advanced or metastatic disease.
* HER2 overexpression defined as HER2 IHC 2+ or 3+.
* Measurable disease according to RECIST 1.1.

Exclusion Criteria:

* Known hypersensitivity to Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection.
* History of receiving any anti-cancer drug/biologic treatment within 4 weeks prior to trial treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate （ORR） | up to 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by investigator | up to 24 months
  Tumor response was assessed by investigator according to RECIST v1.1
Overall Survival(OS) | up to 24 months
  OS was defined as the time from the first study treatment to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peng Z, Liu T, Wei J, Wang A, He Y, Yang L, Zhang X, Fan N, Luo S, Li Z, Gu K, Lu J, Xu J, Fan Q, Xu R, Zhang L, Li E, Sun Y, Yu G, Bai C, Liu Y, Zeng J, Ying J, Liang X, Xu N, Gao C, Shu Y, Ma D, Dai G, Li S, Deng T, Cui Y, Fang J, Ba Y, Shen L. Efficacy and safety of a novel anti-HER2 therapeutic antibody RC48 in patients with HER2-overexpressing, locally advanced or metastatic gastric or gastroesophageal junction cancer: a single-arm phase II study. Cancer Commun (Lond). 2021 Nov;41(11):1173-1182. doi: 10.1002/cac2.12214. Epub 2021 Oct 19. PMID 34665942